CLINICAL TRIAL: NCT05888896
Title: Effect of Foot Reflexology on Preeclampsia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abeer Ali Ahmed Mansour, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: p.t.REC/012/003568
Record Dates: First submitted 2023-05-25; First posted 2023-06-05 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-06

CONDITIONS: Mild Pre-eclampsia
Keywords: Foot reflexology - Preeclampsia - Proteinuria
MeSH Terms: interventions — Methyldopa; Antihypertensive Agents

STUDY DESIGN:
Intervention Model Description: anti-hypertensive drugs and foot reflexology
Who Masked: Participant, Outcomes Assessor
Masking Description: double( Participants, outcomes Assessor)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anti-hypertensive drugs (Experimental): Methyldopa tablets 250 mg will be used oral to reduce hypertension
  Interventions: Other: methyldopa tablets 250mg
- anti-hypertensive drugs+foot reflexology (Experimental): Methyldopa tablets 250 mg and foot reflexology sessions for 8 weeks ( 30 min 2 times per week) will be used to reduce hypertension
  Interventions: Other: methyldopa tablets 250mg + foot reflexology

INTERVENTIONS:
Other: methyldopa tablets 250mg — patients will be taken methyldopa tablets 250mg in the morning orally with a lot of water after breakfast daily and this medication continues for 8 weeks
  Other Names: anti-hypertensive drugs
  Arms: anti-hypertensive drugs
Other: methyldopa tablets 250mg + foot reflexology — patients will receive methyldopa tablets 250mg in oral way once daily per 8 weeks and patients will receive foot reflexology two sessions per week, every session will last for 30 minutes and sessions will last for 8 weeks.
  Other Names: anti-hypertensive drugs+ foot massage
  Arms: anti-hypertensive drugs+foot reflexology

SUMMARY:
the aim of this study to investigate the effect of foot reflexology on mild preeclampsia during pregnancy

DETAILED DESCRIPTION:
Preeclampsia is defined as arterial hypertension identified for the first time after the 20th week associated with proteinuria. It affects 5% to 7% of all pregnant women. It is more common in primigravida women, women with previous early onset preeclampsia, in age greater than 40 years, previous history of preeclampsia, pre-pregnancy obesity, women who become pregnant with donor eggs, embryo donation and donor insemination. It is responsible for over 70 000 maternal deaths and 500 000 fetal deaths worldwide every year. There are many risk factors for it as: Hypertension, diabetes mellitus, proteinuria, obesity, family history, null parity, multiple pregnancies, use of contraception, older women conception (> 40) and thrombotic vascular disease,edema, renal failure, liver failure and hellp syndrome.Complementary therapies such as massage and foot reflexology are used with patients of preeclampsia, it is to normalize the body's function, break down tension, alleviate stress, improve nerve function and blood supply throughout the body. this trial has two groups; one will receive anti-hypertensive drugs and the second will receive anti-hypertensive drugs+foot reflexology sessions for 8 weeks (30 min, 2 session/ week).

ELIGIBILITY:
Inclusion Criteria:

* Their ages were ranged between 20-36 years old.
* Their body mass index was not exceeding 35 kg/m2.
* All women were diagnosed as mild preeclampsia.
* All women were primipara and multipara.

Exclusion Criteria:

* Any fractures in foot.
* Foot ulcer & infection.
* Open skin wound in foot.
* History of stroke.
* Women less than 20 years and more than 36 years.
* BMI more than 35 Kg\m2.
* Severe preeclampsia.

Ages: 20 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant female with preeclampsia
Enrollment: 60 (Estimated)
Dates: Start 2023-06-09 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2023-09-20 (Estimated)

PRIMARY OUTCOMES:
Mean arterial blood pressure | 8 weeks
  the scale that will be used; the Mercury Pressure and Stethoscope; each patient will measured blood pressure before and after treatment

SECONDARY OUTCOMES:
Overall quality of life questionnaire | 8 weeks
  World Health Organization Quality of Life Questionnaire will be used to determine quality of life before and after treatment for all patients
Serum cortisol | 8 weeks
  blood sample will be used to measure level of cortisol before and after treatment
Proteinuria | 8 weeks
  Urine reagent strip devices (dipsticks) will be used to discover it in urine before and after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Abeer Ali Ahmed Mansour, Asyut, Assuit, Egypt